CLINICAL TRIAL: NCT01465438
Title: Can New Imaging- and Biomarkers Improve the Assessment of Disease Activity and Progression and Predict Therapeutic Outcome in Psoriatic Arthritis Patients Receiving Adalimumab?
Brief Title: HUmira in Psoriatic Arthritis
Acronym: HUPSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Copenhagen University Hospital at Herlev (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Professor Mikkel Østergaard, Rheumatologic Research Unit and Department of Rheumatology, Glostrup University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUPSA HUM 05-040; 2006-000004-16 (EudraCT Number)
Record Dates: First submitted 2011-06-16; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-02

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adalimumab (Experimental): Responders at week 24 continue treatment with adalimumab. Non-responders at week 24 stops treatment with adalimumab.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 40 mg every other week
  Other Names: Humira

SUMMARY:
Psoriatic arthritis (PsA) is an inflammatory arthritis associated with psoriasis, which has a estimated prevalence of 0.3 - 1 %. The clinical course varies, but PsA is often a progressive, erosive arthritis causing severe disability and increased mortality.

The biologic treatment infliximab and etanercept have recently been introduced for treatment of PsA and psoriasis, and current data indicate a higher efficacy than with previously available therapies. No clinical trials on adalimumab in PsA are yet published (2005), but preliminary data are encouraging. The improved treatment options have increased the need for sensitive methods for diagnosis, monitoring and prognostication of PsA, so that the efficient therapies can be initiated at the optimal time point and monitored optimally. Ultrasonography (US) and magnetic resonance imaging (MRI) and a number of biomarkers are promising, but not yet sufficiently studied, methods for this.

The hypothesis is that adalimumab will be an effective treatment option for PsA. Novel imaging- and biomarkers can provide additional information, compared to clinical measures and radiography, concerning activity, destructive progression and prediction of therapeutic response in PsA patients receiving adalimumab. The perspective is a potential improvement in diagnosis, monitoring and prognostication of patients with PsA.

ELIGIBILITY:
Inclusion Criteria:

Subject Population: patients with active PsA, fulfilling the following major criteria:

1. Diagnosis of PsA according to Moll and Wright criteria (Moll and Wright,
2. Clinical active disease, defined as >2 (of 76) swollen joints and > 2 (of 78) tender joints
3. Involvement of the hands (Clinical swelling of 1 or more finger joint and/or 1 or more 1 sausage finger)
4. Clinical indication for anti-TNF alpha therapy, according to treating physician
5. Among other issues: Age >18 years; adequate birth control; no contraindications for anti-TNF alpha-therapy, no previous anti-TNF alpha-therapy, no other significant dermatological disorders than psoriasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Modified Psoriatic Arthritis Response criteria (PsARC) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Wiell, MD, PhD, Study Chair — University Hospital, Gentofte, Copenhagen; Inge Juul Sørensen, MD, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre; Michael Sejer Hansen, MD, PhD, Principal Investigator — Copenhagen University Hospital at Herlev; Ole Rintek Madsen, MD, PhD, Principal Investigator — University Hospital, Gentofte, Copenhagen; Ole Slot, MD, Principal Investigator — Glostrup University Hospital, Copenhagen; Susanne J Pedersen, MD, Principal Investigator — Gentofte University Hospital
Locations (1):
- Copenhagen University Hospital, Glostrup, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Poggenborg RP, Wiell C, Boyesen P, Boonen A, Bird P, Pedersen SJ, Sorensen IJ, Madsen OR, Slot O, Moller JM, Hasselquist M, Kubassova O, Ostergaard M. No overall damage progression despite persistent inflammation in adalimumab-treated psoriatic arthritis patients: results from an investigator-initiated 48-week comparative magnetic resonance imaging, computed tomography and radiography trial. Rheumatology (Oxford). 2014 Apr;53(4):746-56. doi: 10.1093/rheumatology/ket426. Epub 2013 Dec 24. PMID 24369412